CLINICAL TRIAL: NCT02088736
Title: Clinical Evaluation of Intraosseous and Intravenous Access for Cardiac Arrest Treatment in Emergency Ambulances In Singapore
Brief Title: Intraosseous vs Intravenous Access for Cardiac Arrest Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Civil Defence Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB 2013/676/C; NMRC/CNIG/1110/2013 (Other: MOH NMRC, Singapore)
Record Dates: First submitted 2014-03-11; First posted 2014-03-17 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Cannula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous and Intraosseous (Active Comparator): 'IV + IO' Intravenous fluids or medications needed and a peripheral IV given 2 attempts or 90 seconds. If IV is unsuccessful, IO will attempt at the Primary site (proximal tibia). If IO is unsuccessful at scene, 2nd attempt can be done in the ambulance. Adrenaline will be delivered as according to protocol.
  Interventions: Device: Intraosseous
- Intravenous (Experimental): Intravenous fluids or medications needed and a peripheral IV given 2 attempts or 90 seconds. If 1st IV is unsuccessful at scene, 2nd IV attempt can be done in the ambulance. Adrenaline will be delivered according to protocol.
  Interventions: Device: Intravenous

INTERVENTIONS:
Device: Intraosseous
  Other Names: EZIO
  Arms: Intravenous and Intraosseous
Device: Intravenous
  Other Names: IV Cannula
  Arms: Intravenous

SUMMARY:
In patients with out-of-hospital cardiac arrest in Singapore, investigators aim to assess the benefit of introducing a resuscitation protocol including the use of intravenous (IV) access and/or intraosseous (IO) vascular access in the pre-hospital setting.

The assumption is that low vascular access rates could be due to difficulty of setting IV cannulas in the field due to certain factors like poor lighting or space constraints. Thus, by introducing a protocol including IO access for difficult IV cases, success rates for vascular access will be higher and this might lead to higher survival rates.

This will be a study comparing 'IV+IO' and 'IV alone' protocols in patients with cardiac arrest managed by Singapore Civil Defence Force (SCDF) emergency ambulance service. The trial will recruit 400 patients over 1 year. Each of the 30 SCDF ambulances will provide both 'IV+IO' and 'IV alone' treatments in 2 consecutive phases of 6-months in order to allow for all ambulance crew a chance to be trained on usage of IO. Currently, IO insertion is the accepted standard of care in Singapore General Hospital, Department of Emergency Medicine.

DETAILED DESCRIPTION:
Primary objectives:

In adult and paediatric patients with Out-of-Hospital Cardiac Arrest (OHCA) in Singapore, investigators aim to evaluate the incremental benefit of introducing a resuscitation protocol including the use of intravenous (IV) access and/or intraosseous (IO) vascular access compared to protocols with only intravenous (IV) access by SCDF paramedics in the pre-hospital setting on the return of spontaneous circulation (ROSC) rates.

Secondary Objective:

* To compare the success rates of vascular access with IV access and/or IO insertion compared to that with intravenous (IV) access alone by SCDF paramedics in the pre-hospital setting.
* To compare the rates of successful 1st dose adrenaline given in the field to cardiac arrest patients in IV+IO and IV groups and whether this translates into a higher survival rate at 30 days.
* To determine the cost benefit of introducing IO access to the emergency ambulance service for OHCA.

Hypothesis:

In adult and paediatric patients with Out-of-Hospital Cardiac Arrest (OHCA) in Singapore, the hypothesis is that low vascular access rates could be due to difficulty of setting IV cannulas in the field due to certain factors like poor lighting or space constraints. Thus, by introducing a protocol including IO access for difficult IV cases, success rates for vascular access will be higher and this might lead to a higher ROSC and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest (medical or traumatic)
* Intravenous fluids or medications needed

Exclusion Criteria:

* Adult needle (weight ≥ 40 kg)
* Paediatric needle (weight 3 - 39 kg)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1103 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Any Return of Spontaneous Circulation Rate (ROSC) | At scene to hospital (about 2 hours)
  Any ROSC including transient or intermittent during pre- or in-hospital

SECONDARY OUTCOMES:
Insertion success rate | 90 secs
Number of patients administered 1st dose | 90 secs
Survival outcome | up to 30 days
Time taken for 1st dose of adrenaline given | 90 secs

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Boon Kiat Tan, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore Civil Defence Force, Singapore, Singapore